CLINICAL TRIAL: NCT00529035
Title: A Phase I Study of Ultra-Low Dose Subcutaneous Interleukin-2 (IL-2) for Treatment of Refractory Chronic Graft Versus Host Disease
Brief Title: Ultra-Low Dose Interleukin-2 for Refractory Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Novartis (Industry)
Responsible Party: Principal Investigator, John Koreth, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-083
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Graft Versus Host Disease
Keywords: Chronic GVHD; Steroid refractory GVHD; allogeneic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interleukin-2 (Experimental): Interleukin-2 (IL-2) will be given daily through an injection under the skin for a period of 8 weeks. To determine the highest safest dose of IL-2, the dose participants receive will increase as lower doses are determined to be safe. There will be three dose levels:
  Dose Level -A 0.3 x 106 (IU/m2/d) Dose Level -B 1 x 106 (IU/m2/d) Dose Level-C 3 x 106 (IU/m2/d)
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — Dose will vary depending upon when participant enters the trial: Given as a daily injection under the skin for 8 weeks.
  Other Names: IL-2

SUMMARY:
The purpose of this research study is to determine the safety of IL-2 and the highest dose of this drug that can be given safely to people with chronic graft versus host disease (GVHD). Chronic GVHD is a medical condition that may occur after patients receive a bone marrow, stem cell or cord blood transplant. The donor's immune system may recognize their body (the host) as foreign and attempt to "reject" it. Traditional standard therapy to treat chronic GVHD is prednisone (steroids). Treatment options are limited, and it is thought that IL-2 may help to control chronic GVHD.

DETAILED DESCRIPTION:
* IL-2 will be given daily through an injection under the skin for a period of 8 weeks. To determine the highest safest dose of IL-2, the dose participants receive will increase as lower doses are determined to be safe. There will be three dose levels.
* Participants will be seen periodically while they are receiving IL-2. Physical exams and blood tests will be performed weekly for the first two weeks and then every other week until week 8.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of allogeneic stem cell transplantation with myeloablative or non-myeloablative conditioning regimens
* Patients must be at least 180 days from the allogeneic stem cell transplantation procedure
* Steroid refractory cGVHD, defined as having persistent symptoms and signs of GVHD despite the use of prednisone for at least 4 weeks in the preceding 12 months without complete resolution of signs and symptoms.
* Stable dose of corticosteroids for 4 weeks prior to enrollment
* No addition or subtraction of other immunosuppressive medications for 4 weeks prior to enrollment.
* Adequate bone marrow, renal and hepatic function as outlined in the protocol
* 18 years of age or older
* ECOG Performance Status of 0-2

Exclusion Criteria:

* Ongoing prednisone requirement > 1mg/kg/day (or equivalent)
* Exposure to any new immunosuppressive medication in the 4 weeks prior to enrollment
* Concurrent ECP therapy within 4 weeks prior to enrollment
* Post-transplant exposure to any novel immunosuppressive medication within 100 days prior to enrollment
* Donor lymphocyte infusion within 100 days prior to IL-2 therapy
* Active malignant disease relapse
* Active, uncontrolled infection
* Positive serologic test for Hepatitis B or a positive serologic or nucleic acid test for Hepatitis C
* HIV seropositivity
* Life expectancy < 3 months
* Pregnancy or lactation
* Inability to comply with IL-2 treatment regimen
* Uncontrolled cardiac angina or symptomatic congestive heart failure
* Organ transplant (allograft) recipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-08; Primary Completion 2011-06 (Actual); Study Completion 2020-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Koreth, MBBS, D.Phil, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

REFERENCES:
- [Result] Koreth J, Matsuoka K, Kim HT, McDonough SM, Bindra B, Alyea EP 3rd, Armand P, Cutler C, Ho VT, Treister NS, Bienfang DC, Prasad S, Tzachanis D, Joyce RM, Avigan DE, Antin JH, Ritz J, Soiffer RJ. Interleukin-2 and regulatory T cells in graft-versus-host disease. N Engl J Med. 2011 Dec 1;365(22):2055-66. doi: 10.1056/NEJMoa1108188. PMID 22129252

RESULTS

PARTICIPANT FLOW:
Groups:
- Ultra-low Dose Interleukin-2: Daily subcutaneous administration of Interleukin-2 evaluated at three dose levels:
  Dose level A: 0.3 x 10^6 IU/m^2/day Dose level B: 1.0 x 10^6 IU/m^2/day Dose level C: 3.0 x 10^6 IU/M^2/day
Period: Overall Study
Arm/Group | Ultra-low Dose Interleukin-2
Started | 29 (29 enrolled)
Completed | 28 (28 evaluable, 1 patient withdrew participation and was not evaluable)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Interleukin-2 (IL-2) will be given daily through an injection under the skin for a period of 8 weeks. To determine the highest safest dose of IL-2, the dose participants receive will increase as lower doses are determined to be safe. There will be three dose levels:
  Dose Level -A 0.3 x 106 (IU/m2/d) Dose Level -B 1 x 106 (IU/m2/d) Dose Level-C 3 x 106 (IU/m2/d)
Arm/Group | Group 1
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose and Toxicity Profile of an 8 Week Course of IL-2 in Patients With cGVHD and an Inadequate Response to Steroids.
Description: Three dose levels were evaluated to determine the maximally tolerated dose (MTD):
  Dose level A: 0.3 x 10^6 IU/m^2/day Dose level B: 1.0 x 10^6 IU/m^2/day Dose level C: 3.0 x 10^6 IU/m^2/day Once the MTD (dose level B) was established, an additional 10 participants were enrolled at this dose.
Time Frame: Participants were assessed for toxicities at mandatory study follow-up visits during the 8 week course of study therapy and four weeks post therapy
Population: One participant terminated therapy early and was not evaluable for this outcome measure.
Measure: Number; unit: million IU/m2/day
Arm/Group | Ultra-low Dose IL-2 MTD
Number analyzed (Participants) | 28
million IU/m2/day | 1

2. Secondary Outcome: The Number of Participants Who Tolerated at Least 6 Weeks of Subcutaneous Low Dose IL-2.
Description: Feasibility: the number of participants who tolerated at least 6 weeks of therapy, and were thus evaluable for response. Efficacy: chronic GVHD response per NIH consensus criteria in evaluable patients.
  A complete response was defined as resolution of all reversible chronic GVHD-associated manifestations, a partial response as an improvement of 50% or more on the organ-specific chronic GVHD scale without progression at other organs or sites, progressive disease as an increase of 25% or more on the organ specific chronic GVHD scale, and stable disease as an improvement of less than 50% or increase of less than 25%. Please refer to the Supplementary Appendix in our published report (Koreth et al, NEJM 2011) for further details.
Time Frame: Participants were assessed for toxicities at mandatory study follow-up visits during the 8 week course of study therapy and four weeks post therapy. cGVHD was assessed at Weeks 8 and 12
Population: Participants were evaluable for response and considered meeting the feasibility endpoint if they completed at least 6 weeks of treatment. Participants who had a partial response or complete response in cGVHD to treatment were considered to meet the efficacy endpoint.
Measure: Number; unit: participants
Arm/Group | Ultra-low Dose Interleukin-2
Number analyzed (Participants) | 28
participants
  Feasibility | 23
  Efficacy | 12

3. Secondary Outcome: CD3+T, CD4+T (Including Regulatory CD4+T Cells (Treg) and Conventional CD4+T Cells (Tcon)), CD8+T, NK, NKT and B Cell Counts.
Description: Changes in the above immune cell populations (CD3+T, CD4+T (including CD4+Treg and CD4+Tcon), CD8+T, NK, NKT and B cell counts were measured at study appointments during the 8-week IL-2 treatment and four weeks post study therapy.
  All study participants (n=28) with a sample available were reported in the data table.
  Immune outcome data cannot be meaningfully rendered in the template provided, owing to complexity. The tables below only represent a general overview of the data. Please refer to figure 2 in our published report (Koreth et al, NEJM 2011).
Time Frame: Immunological samples taken at study appointments during the 12 week protocol schedule
Population: Participants were evaluated for regulatory T cell (Treg) expansion and other immune-cell changes while on low-dose IL-2 therapy. Participants had blood samples drawn at study appointments during the 12 week protocol schedule. Please note that for NK and NKT cell counts, only 18 participants samples were analyzed.
Measure: Median (Inter-Quartile Range); unit: cells/cubic millimeter
Groups:
- Median Absolute Cell Counts at Baseline: Immune-cell counts before the start of IL-2 therapy
- Median Absolute Cell Counts at Week 8: Immune-cell counts after 8 weeks of IL-2 therapy
- Median Absolute Cell Count at Week 12: Immune-cell counts after a 4 weeks off IL-2 per protocol
Arm/Group | Median Absolute Cell Counts at Baseline | Median Absolute Cell Counts at Week 8 | Median Absolute Cell Count at Week 12
Number analyzed (Participants) | 22 | 19 | 15
cells/cubic millimeter
  Treg cell count | 17 [6 to 35] | 101 [43 to 236] | 32 [11 to 92]
  Tcon cell count | 206 [131 to 412] | 270 [110 to 678] | 209 [153 to 550]
  CD8+ T cell count | 210 [113 to 419] | 202 [74 to 418] | 187 [55 to 502]
  Natural Killer (NK) cell count | 158 [94 to 250] | 362 [170 to 570] | 203 [132 to 311]
  NKT cell count | 28 [10 to 46] | 31 [18 to 53] | 22 [10 to 38]

4. Secondary Outcome: Treg Cell:Tcon Cell Ratio
Description: Changes in the ratio of the CD4+ regulatory T cell (Treg) and CD4+ conventional T cell (Tcon) counts were measured at study appointments during the 8-week IL-2 treatment and four weeks post study therapy.
  All study participants (n=28) with a sample available were reported in the data table.
  Immune outcome data cannot be meaningfully rendered in the template provided, owing to complexity. The tables below only represent a general overview of the data. Please refer to figure 2 in our published report (Koreth et al, NEJM 2011).
Time Frame: Immunological samples taken at study appointments during the 12 week protocol schedule
Population: Participants were evaluated for changes to the ratio of regulatory T cell (Treg) and conventional T cell (Tcon) counts while on IL-2 therapy. Participants had blood samples drawn at study appointments during the 12 week protocol schedule to analyze the immunological effects of low-dose IL-2 therapy.
Measure: Median (Inter-Quartile Range); unit: ratio
Groups:
- Median Treg:Tcon Ratio at Baseline: Immune-cell ratio before the start of IL-2 therapy
- Median Treg:Tcon Ratio at Week 8: Immune-cell ratio after 8 weeks of IL-2 therapy
- Median Treg:Tcon Ratio at Week 12: Immune-cell ratio after a 4 weeks off IL-2 per protocol
Arm/Group | Median Treg:Tcon Ratio at Baseline | Median Treg:Tcon Ratio at Week 8 | Median Treg:Tcon Ratio at Week 12
Number analyzed (Participants) | 22 | 19 | 15
ratio | 0.07 [0.05 to 0.12] | 0.4 [0.24 to 0.71] | 0.14 [0.09 to 0.22]

ADVERSE EVENTS:
Time Frame: 12 weeks. For patients who continued on extended-duration therapy, adverse events were reported as long as they received treatment.
Groups:
- Ultra-low Dose Interleukin-2: Interleukin-2 (IL-2) will be given daily through an injection under the skin for a period of 8 weeks. To determine the highest safest dose of IL-2, the dose participants receive will increase as lower doses are determined to be safe. There will be three dose levels:
  Dose Level -A 0.3 x 106 (IU/m2/d) Dose Level -B 1 x 106 (IU/m2/d) Dose Level-C 3 x 106 (IU/m2/d)
Arm/Group | Ultra-low Dose Interleukin-2
Serious Adverse Events (participants affected / at risk) | 9/29
Other Adverse Events (participants affected / at risk) | 4/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultra-low Dose Interleukin-2 (N=29)
Thrombotic microangiopathy with renal failure (Blood and lymphatic system disorders) | 2 (2)
MRSA Pneumonia (Infections and infestations) | 1 (1) — Subject with MRSA pneumonia documented prior to start of study treatment had recrudescent MRSA pneumonia at week 7.
MRSA furuncle (Infections and infestations) | 1 (1) — MRSA furuncle preceded start of study treatment.
Hemophilius influenza type B bacteremia (Infections and infestations) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) — On subject experienced a fatal acute myocardial infarction 70 days after coming off-treatment (unrelated to study treatment). Another subject, with known coronary artery disease, had a myocardial infarction at 2 weeks off-treatment.
Injection site induration (General disorders) | 2 (2) — 2 subjects experienced reversible injection site induration reactions.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultra-low Dose Interleukin-2 (N=29)
Constitutional symptoms (General disorders) | 2 (2) — 2 subjects had low-grade constitutional symptoms (fever, malaise, arthralgia)
Renal dysfunction (mild) (Renal and urinary disorders) | 1 (1)
Thrombocytopenia (mild) (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes